CLINICAL TRIAL: NCT02197598
Title: Exploratory, Interventional, Open-label, Fixed-dose Study With Selincro® As-needed Use, in Alcohol Dependent Patients With Liver Impairment
Brief Title: Treatment of Patients Suffering of Alcohol Dependence and Impaired Liver Function With Selincro® As-needed Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15871A; 2014-000413-31 (EudraCT Number)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Alcohol Dependence
Keywords: nalmefene, alcohol consumption, liver effects
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selincro® (nalmefene) 18 mg, tablets (Experimental): One tablet orally for 12 weeks on days when the patient perceives a risk of drinking alcohol, preferably 1-2 hours prior to the anticipated risk of drinking.
  Interventions: Drug: nalmefene

INTERVENTIONS:
Drug: nalmefene
  Other Names: Selincro®

SUMMARY:
The purpose of this study is to explore the treatment effects of Selincro in alcohol dependent patients with liver impairment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has alcohol dependence, diagnosed at screening according to DSM-IV-TR™
* The patient has had an average alcohol consumption at, at least, a high drinking risk level (that is >60 g of alcohol/day for men and >40 g of alcohol/day for women) in the 4 weeks preceding the Screening Visit and in the period between the Screening and Inclusion Visits (that is, in the Screening Period)
* The patient has liver impairment defined by elevated liver stiffness and elevated liver enzymes at the Screening Visit (both criteria have to be fulfilled): liver stiffness (LS) as measured by Fibroscan >6 kPa, elevated transaminases (AST or ALT). Transaminase levels up to 5 times the upper limit of the reference range and γGT levels up to 10 times the upper limit of the reference range are allowed. At the discretion of the investigator, transaminase levels >5 times the upper limit of the reference range and γGT >10 times the upper limit of the reference range can be allowed if considered habitual for the patient, either confirmed by patient records or a repeat measurement during the Screening Period
* The patient has a breath alcohol concentration (BrAC) <0.02% at the Screening Visit.
* The patient provides a stable address and telephone number
* The patient is a man or woman, aged ≥ 18 years
* The patient has BMI≤30 kg/m2

Exclusion Criteria:

* The patient has any psychiatric disorder or Axis I disorder (DSM-IV-TR™ criteria), established as the primary diagnosis, other than alcohol dependence assessed using the Mini International Neuropsychiatric Interview (MINI) or another diagnostic interview , that in any way will interfere with the ability of the patient to take part in the study
* The patient has reported current use of, or has been tested positive for, drugs of abuse (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates)
* The patient has severe liver impairment classified with a Child-Pugh Score C
* The patient has one or more clinical laboratory test values outside the reference range, based on the blood and urine samples taken at the Screening Visit, that are of potential risk to the patient's safety, or the patient has: Severe renal impairment (eGFR <30 mL/min per 1.73 m2), and/or Hypercholesterolemia with serum cholesterol levels > 300 mg/dL, (>7,758 mmol/L), and/or bilirubin > 3 mg/dL (50 μmol/L)
* The patient has had <6 heavy drinking days (HDDs, defined by the European Medicines Agency as a day with an alcohol consumption >60 g for men or >40 g for women) in the 4 weeks preceding the Screening Visit
* The patient has >5 consecutive abstinence days in the 4 weeks preceding the Screening Visit
* The patient has a recent history of acute alcohol withdrawal syndrome (including hallucinations, seizures, or delirium tremens)

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of heavy drinking days per month (HDDs) (days/month) | Baseline to months 1, 2 and 3
Change from baseline in the number of HDDs per week (days/week) | Baseline to weeks 1 and 2
Change from baseline in total alcohol consumption (TAC) (g alcohol/day) | Baseline to months 1, 2 and 3
Change from baseline in TAC (g alcohol/day) | Baseline to weeks 1 and 2
Response Shift Drinking Risk Level (RSDRL) | Baseline to month 3
  Defined as a downward shift from baseline in drinking risk level (DRL); for patients with a very high DRL at baseline, a shift to medium DRL or lower; for patients with a high DRL at baseline, a shift to low DRL or below
Response Low Drinking Risk Level (RLDRL) | Baseline to month 3
  Defined as a downward shift from baseline in DRL to low DRL or below
Response defined as ≥70% reduction in TAC | Baseline to month 3
Response defined as 0 to 4 HDDs (days/month) | Month 3
Clinical Global Impression, global improvement (CGI-I). | Weeks 4 and 12
Change from baseline in Clinical Global Impression, Severity of illness (CGI-S) | Baseline to weeks 4 and 12
Change in the Short-Form 36-Item Health Survey (SF-36) | Baseline to week 12
Change in liver stiffness | Baseline to weeks 1,2 4 and 12
Category shift in fibrosis stage | Baseline to weeks 1,2 4, and 12
Change in transaminases and γ-glutamyl transferase (γGT) | Baseline to weeks 1,2,4,8, and 12
Change in bilirubin, albumin, and International Normalized Ratio (INR) | Baseline to weeks 1,2,4,8, and 12
Number of adverse events | Screening to week 14

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (3):
- Germany (3):
  - DE001, Heidelberg
  - DE002, Mannheim
  - Optuminisight, München

REFERENCES:
- Available data/document: EMA EudraCT Results: 2014-000413-31 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-000413-31/results